CLINICAL TRIAL: NCT00993863
Title: A Randomized, Single-Dose, Double-Blind, Active- and Placebo-Controlled Study of ADL5859 for the Treatment of Pain After Surgical Removal of Impacted Third Molars
Brief Title: Analgesic Efficacy and Safety of ADL5859 in Subjects With Acute Dental Pain After Third Molar Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Senior Medical Director, Clinical Research, Adolor Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 33CL230; 33CL230
Record Dates: First submitted 2009-10-09; First posted 2009-10-14 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2009-10

CONDITIONS: Acute Pain
Keywords: delta opioid agonist; dental pain
MeSH Terms: conditions — Acute Pain; Toothache | interventions — N,N-diethyl-4-(5-hydroxyspiro(chromene-2,4'-piperidine)-4-yl)benzamide; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- ADL5859 30 mg (Experimental)
  Interventions: Drug: ADL5859 30 mg
- ADL5859 100 mg (Experimental)
  Interventions: Drug: ADL5859 100 mg
- ADL5859 200 mg (Experimental)
  Interventions: Drug: ADL5859 200 mg
- ibuprofen 400 mg (Active Comparator)
  Interventions: Drug: ibuprofen 400 mg

INTERVENTIONS:
Drug: Placebo — single dose
  Arms: Placebo
Drug: ADL5859 30 mg — single dose
  Arms: ADL5859 30 mg
Drug: ADL5859 100 mg — single dose
  Arms: ADL5859 100 mg
Drug: ADL5859 200 mg — single dose
  Arms: ADL5859 200 mg
Drug: ibuprofen 400 mg — single dose
  Other Names: Advil
  Arms: ibuprofen 400 mg

SUMMARY:
The objective of this study is to evaluate the analgesic efficacy and safety of ADL5859 compared with placebo and an active control (ibuprofen) in subjects with acute dental pain after third molar extraction.

ELIGIBILITY:
Key Inclusion Criteria:

* have 2 or more 3rd molars requiring extraction, including at least 1 partially or completely bone-impacted mandibular molar
* experience moderate to severe pain intensity as measured by the Numeric Pain Rating Scale (NPRS) (score ≥ 5) within 6 hours after surgery
* for male subjects, be surgically sterile or agree to use an appropriate method of contraception or have a sexual partner who is surgically sterile or using an insertable, injectable, transdermal, or combination oral contraceptive
* for female subjects, be using contraceptives, be postmenopausal, or have undergone hysterectomy or tubal ligation
* be able to take oral study medications

Key Exclusion Criteria:

* have positive results either on the urine screening tests for opiates, tetrahydrocannabinol,cocaine, amphetamines, barbiturates, benzodiazepines, phencyclidine, or propoxyphene or on the alcohol breathalyzer test
* have a history of alcoholism or drug addiction or abuse within 5 years before dosing with study medication
* have a history of chronic use (defined as daily use for > 2 weeks) of glucocorticoids,nonsteroidal anti-inflammatory drugs, or opiates for any condition within 6 months of study medication administration
* have a known allergy or history of significant reaction to any of the known treatment medications (ADL5859-like compounds or ibuprofen) or rescue pain medication (acetaminophen)
* have significant renal or hepatic disease, as indicated by clinical laboratory assessment
* have a known history of epilepsy or seizure disorder, including history of febrile seizure, or any other medical or psychiatric condition that, in the judgment of the investigator, would put the subject at risk while in the study, could influence the results of the study, or could negatively affect the subject's ability to participate in the study
* have a history or evidence of orthostatic hypotension at screening have a history of significant head trauma (head injury with loss of consciousness)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2007-06; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Total pain relief 0-4 hours after study medication | 4 hours after study medication

CONTACTS AND LOCATIONS:
Locations (1):
- SCIREX Research Center, Austin, Texas, United States